CLINICAL TRIAL: NCT07323017
Title: Electrochemotherapy in Musculoskeletal Tumors: A Quantitative Assessment of Tumor Size Variations and Treatment-related Pain Reduction.
Brief Title: Electrochemotherapy in Musculoskeletal Tumors
Status: Active, not recruiting | Type: Observational
Sponsor: Costantino Errani (Other)
Responsible Party: Sponsor-Investigator, Costantino Errani, Principal Investigator, Istituto Ortopedico Rizzoli
Organization: Istituto Ortopedico Rizzoli (Other)
Other Study IDs: ELECTRO
Record Dates: First submitted 2025-12-10; First posted 2026-01-07 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Bone Tumors
MeSH Terms: conditions — Bone Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study involves the enrollment of patients over 2 years of age with a diagnosis of musculoskeletal tumors and an indication for electrochemotherapy, treated at the Rizzoli Orthopaedic Institute in Bologna and followed during outpatient follow-up. Data will be collected from medical records, outpatient reports, and imaging studies including CT, X-ray, MRI, and/or PET.

For the retrospective part of the study, patients treated at the Rizzoli Orthopaedic Institute from 01/01/2024 to the date of approval of this study will be included. For the prospective part, patients meeting the inclusion criteria and treated from the study start date until 31/12/2030 will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes with a histological diagnosis of a primary musculoskeletal tumor, either benign or malignant, located outside the abdominal cavity (trunk and limbs)
* Indication for electrochemotherapy due to one of the following conditions:

  1. Clinical conditions contraindicating surgery
  2. Tumor not surgically resectable
* Patients treated with electrochemotherapy at the Rizzoli Orthopaedic Institute:

  1. From 01/01/2024 to the date of study approval for the retrospective phase
  2. From the date of study approval to 12/31/2030 for the prospective phase
* Retrospectively treated patients with a minimum follow-up of at least 3 months
* Age ≥ 2 years at the time of treatment
* Availability of clinical and instrumental data

Exclusion Criteria:

• Failure to meet at least one of the inclusion criteria

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include patients older than 2 years with a diagnosis of musculoskeletal tumors who are indicated for electrochemotherapy, treated at the Rizzoli Orthopaedic Institute in Bologna and followed during outpatient follow-up. Data will be collected from medical records, outpatient reports, and imaging studies (CT, X-ray, MRI, and/or PET).
  The retrospective part will include patients treated at the Rizzoli Orthopaedic Institute from January 1, 2024, to the date of study approval.
  The prospective part will enroll patients meeting the inclusion criteria who will be treated from the study start date until December 31, 2030.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2030-12-30 (Estimated); Study Completion 2032-06-30 (Estimated)

PRIMARY OUTCOMES:
Tumor size will be assessed using CT, MRI, X-ray, and/or PET imaging. Tumor size will be defined as the longest diameter of the target lesion (mm). | 3, 6, and 12 months after electrochemotherapy

SECONDARY OUTCOMES:
Change from baseline in pain intensity measured by the Visual Analog Scale (VAS), ranging from 0 to 10, where higher scores indicate worse pain, at 3, 6, and 12 months after electrochemotherapy.Number of participants with treatment-related adverse events | 3, 6, and 12 months after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Istituto Ortopedico Rizzoli, Bologna, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Campanacci L, Cevolani L, De Terlizzi F, Saenz L, Ali N, Bianchi G, Donati DM. Electrochemotherapy Is Effective in the Treatment of Bone Metastases. Curr Oncol. 2022 Mar 4;29(3):1672-1682. doi: 10.3390/curroncol29030139. PMID 35323339
- [Result] Cevolani L, Campanacci L, Staals EL, Dozza B, Bianchi G, De Terlizzi F, Donati DM. Is the association of electrochemotherapy and bone fixation rational in patients with bone metastasis? J Surg Oncol. 2023 Jul;128(1):125-133. doi: 10.1002/jso.27247. Epub 2023 Mar 26. PMID 36966436